CLINICAL TRIAL: NCT01717079
Title: Effect of Transcranial Magnetic Stimulation on Disturbance of Body Shape Perception in Patients With Anorexia Nervosa
Brief Title: rTMS and Body Shape Perception
Acronym: STIMOREX
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Protocol stopped for safety reason
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2011/122/HP
Record Dates: First submitted 2012-09-24; First posted 2012-10-30 (Estimated); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Effective arm (Active Comparator): Effective coil
  Interventions: Procedure: rTMS
- Placebo arm (Placebo Comparator): Placebo coil
  Interventions: Procedure: Sham rTMS

INTERVENTIONS:
Procedure: Sham rTMS — 120 pulses 0.2Hz
  Arms: Placebo arm
Procedure: rTMS — 120 pulses 0.2Hz
  Arms: Effective arm

SUMMARY:
Anorexia nervosa (AN) is a frequent, potentially life-threatening eating disorder characterized by a resistance to maintaining body weight at or above a minimally normal weight for age and height, an intense fear of weight gain or being "fat" even though underweight, a loss of menstrual periods in girls and women post-puberty and a disturbance in the experience of body weight or shape. Body weight and shape dissatisfaction is linked to the development, maintenance and relapse of AN. Neuroimaging studies have shown that the inferior parietal cortex is involved in body image perception and less activated in patients with AN compared with healthy subjects. Repetitive transcranial magnetic stimulation (rTMS) is used to modulate cortical excitability, and particularly to increase excitability with high-frequency rTMS. The aim of this study was to investigate the effect of "excitatory" high-frequency rTMS over the "hypoactive" inferior parietal cortex of 54 patients with AN.

This randomized, double-blind, placebo-controlled study will compare effective rTMS (2000 ten-Hz stimulations per session, applied at 90% of the resting motor threshold, with 10 sessions in two weeks) versus placebo rTMS.

Assessments will be performed before rTMS and after the last rTMS session (immediately after, at 15 days and three months). The principal criteria for judgement is a body image satisfaction scale (Boby Shape Questionnaire, BSQ-34). The secondary criteria for judgement are eating behaviour scales (Eating Attitude Test, EAT-40; Bulimia test, BULIT and Eating Disorders Inventory, EDI-2), the Hamilton depression rating scale and Hamilton anxiety rating scale, a quality of life scale (Short-Form Health Survey, SF-36), a body composition analysis using a Dual-energy X-ray absorptiometry and the alpha-MSH autoantibodies levels (biomarker for eating disorders recently described).

Inferior parietal cortex rTMS could not only improve body image perception, but also help in the treatment of eating disorders, allowing weight gain with a decreased anxiety and improving patients' quality of life. Also positive results could have direct therapeutic implications with the possibility to complete regular rTMS sessions, or to implant extradural electrodes for chronic parietal cortex stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age above 18
* Restrictive anorexia nervosa with a disease duration more than one year and less than three years.
* Body Mass Index below 16
* Patient receiving or having received optimal treatment for anorexia nervosa
* Right-handed
* Normal blood ionogramme
* Previous stable antidepressor treatment for one month and no expected modification in the three following months
* Patients arriving by car with someone else or by public transportation

Exclusion Criteria:

* Pregnancy
* Contraindication to transcranial magnetic stimulation i.e. pace-maker, cardiac valve protheses, metallic protheses etc.
* History of epileptic seizure
* Cerebral lesion of any etiology (post-traumatic, tumoral, vascular etc.)
* History of previous rTMS

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
BSQ-34 scale (Body Shape Questionnaire) | Just after rTMS

SECONDARY OUTCOMES:
EAT-40 scale (eating attitude test) | Before rTMS, just after rTMS, 15 days after rTMS and 3 months after rTMS
BULIT scale (bulimia test) | Before rTMS, just after rTMS, 15 days after rTMS and 3 months after rTMS
EDI-2 scale (eating disorder inventory) | Before rTMS, just after rTMS, 15 days after rTMS and 3 months after rTMS
Hamilton scale | Before rTMS, just after rTMS, 15 days after rTMS and 3 months after rTMSBefore rTMS, just after rTMS, 15 days after rTMS and 3 months after rTMS
Quality of Life Scale, MOS 36 Item Short-Form Health Survey or SF-36 | Before rTMS, just after rTMS, 15 days after rTMS and 3 months after rTMS
The body mass index | Before rTMS, just after rTMS, 15 days after rTMS and 3 months after rTMS
body composition analysis using dual energy X-ray absorptiometry | Before rTMS and 3 months after rTMS
autoantibodies against alpha-melanocyte stimulating hormone | Before rTMS, just after rTMS, 15 days after rTMS and 3 months after rTMS
The adverse effects | After rTMS
Weight | Before rTMS, just after rTMS, 15 days after rTMS and 3 months after rTMS
BSQ-34 scale (Body Shape Questionnaire) | Before rTMS, 15 days after rTMS and 3 months after rTMS

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie CHASTAN, MD, Principal Investigator — UH Rouen
Locations (1):
- Rouen University Hospital, Rouen, France